CLINICAL TRIAL: NCT00746486
Title: Double-blind, Randomised, Placebo-controlled, Multi-centre Phase III Clinical Study Comparing the Combination of Ursodeoxycholic Acid Capsules Plus Budesonide Capsules to Ursodeoxycholic Acid Capsules Plus Placebo in the Treatment of Primary Biliary Cirrhosis
Brief Title: Ursodeoxycholic Acid Plus Budesonide Versus Ursodeoxycholic Acid Alone in Primary Biliary Cirrhosis (PBC)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study stopped based on the recommendation of the IDMC after a planned Interim Analysis
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUC-56/PBC; 2007-004040-70
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Primary Biliary Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): One budesonide 3 mg capsule TD or one budesonide 3 mg capsule BD and 12-16 mg ursodeoxycholic acid/kg BW/d
  Interventions: Drug: budesonide
- B (Active Comparator): One placebo capsule TD or One placebo capsule BD and 12-16 mg ursodeoxycholic acid/kg BW/d
  Interventions: Drug: budesonide placebo

INTERVENTIONS:
Drug: budesonide — One budesonide 3 mg capsule TD or one budesonide 3 mg capsule BD and 12-16 mg ursodeoxycholic acid/kg BW/d for 3 years
  Arms: A
Drug: budesonide placebo — One placebo capsule TD or One placebo capsule BD and 12-16 mg ursodeoxycholic acid/kg BW/d for 3 years
  Arms: B

SUMMARY:
The study is aimed to compare the efficacy and tolerability of a combination therapy with ursodeoxycholic acid (12-16 mg/kg body weight (BW)/d) plus budesonide (9 mg/d) vs. ursodeoxycholic acid (12-16 mg/kg BW/d) plus placebo in the treatment of PBC. Depending on ALT values 6 mg/d budesonide are allowed. The study population will be patients with PBC at risk for disease progression. It is assumed that the combination therapy will result in a decrease of treatment failures after 3 years of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Age ≥ 18 years
3. UDCA treatment for at least 6 months prior to inclusion
4. Liver biopsy compatible with PBC
5. Liver biopsy performed within the last 6 months prior to inclusion
6. PBC patients at risk of disease progression based on one or more of the following criteria:

   * Serum alkaline phosphatase ≥ 3 times the upper limit of normal at any time since diagnosis of PBC and ALT ≥ 2 times upper limit of normal or
   * Total Bilirubin ≥ 1.0 mg/dl (≥ 17 µmol/L) or
   * Moderate to severe periportal or periseptal lymphocytic interface hepatitis or
   * Periportal and portal fibrosis with numerous septa (Ludwig stage III) without cirrhosis
7. Type 2 anti-mitochondrial antibodies > 1:40 by direct immunofluorescence
8. Women of child-bearing potential have to apply appropriate contraceptive methods, e.g., hormonal contraception, intrauterine device (IUD), double-barrier method of contraception (e.g., use of a condom and spermicide), partner has undergone vasectomy and subject is in monogamous relationship. The investigator is responsible for determining whether the subject has adequate birth control for study participation

Exclusion Criteria:

1. Histologically proven cirrhosis
2. Positive Hepatitis B or C serology
3. Positive HIV serology
4. Primary Sclerosing Cholangitis
5. Wilson's-Disease
6. Celiac Disease (blood tests and/or oesophago-gastro-duodenoscopy with histological examination to be performed)
7. α1-anti-Trypsin-deficiency
8. Haemochromatosis
9. Autoimmune-Hepatitis (AIH; defined by an Alvarez score > 15 without treatment or ≥ 17 with treatment); Note: PBC/AIH overlap disease, treated insufficiently with UDCA monotherapy may be enrolled
10. Treatment with any of the following drugs within the last 3 months prior to inclusion: colchicine, corticosteroids, azathioprine or other immunosuppressive drugs (e.g. cyclosporine, methotrexate), chlorambucil, D-penicillamine, fibrates, or antihyperlipidemic drugs
11. Treatment with ketoconazole or other CYP3A inhibitors within the last 4 weeks before baseline; rifampicin (up to 600 mg/d) is allowed to treat pruritus until baseline
12. Sonographic or endoscopic signs of portal hypertension
13. Ascites or history of ascites
14. Hepatic encephalopathy or history of hepatic encephalopathy
15. Total bilirubin > 3.0 mg/dl (> 50 µmol/L)
16. Albumin < 36 g/L
17. Prothrombin ratio < 70%
18. Platelet count < 135.000/mm3
19. Osteoporosis proven by bone densitometry
20. Diabetes mellitus, defined as B-Glucose > 125 mg/dl on an empty stomach (even when controlled)
21. Hypertension, defined as persistent raised blood pressure > 140/90 mmHg
22. Suspected non-compliance of the patient (suspected difficulties to comply with the study period of 36 months)
23. Severe co-morbidity substantially reducing life expectancy
24. Known intolerance/hypersensitivity/resistance to study drugs or drugs of similar chemical structure or pharmacological profile
25. Existing or intended pregnancy or breast-feeding
26. Participation in another clinical trial within the last 30 days, simultaneous participation in another clinical trial, or previous participation in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-02; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Rate of patients without treatment failure after 3 years of treatment | 3 years, LOCF

SECONDARY OUTCOMES:
course of pruritus | 3 years, LOCF
course of fatigue | 3 years, LOCF
course of Mayo Risk score | 3 years, LOCF
bone mineral density | 3 years, LOCF

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Poupon, Professor, Principal Investigator — Hôpital Saint-Antoine, 75571 Paris, France
Locations (2):
- Hôpital Saint-Antoine, Paris, France
- Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Hirschfield GM, Beuers U, Kupcinskas L, Ott P, Bergquist A, Farkkila M, Manns MP, Pares A, Spengler U, Stiess M, Greinwald R, Prols M, Wendum D, Drebber U, Poupon R. A placebo-controlled randomised trial of budesonide for PBC following an insufficient response to UDCA. J Hepatol. 2021 Feb;74(2):321-329. doi: 10.1016/j.jhep.2020.09.011. Epub 2020 Sep 17. PMID 32950590
- [Derived] Mousa HS, Lleo A, Invernizzi P, Bowlus CL, Gershwin ME. Advances in pharmacotherapy for primary biliary cirrhosis. Expert Opin Pharmacother. 2015 Apr;16(5):633-43. doi: 10.1517/14656566.2015.998650. Epub 2014 Dec 29. PMID 25543678